CLINICAL TRIAL: NCT02231749
Title: A Phase 3, Randomized, Open-Label Study of Nivolumab Combined With Ipilimumab Versus Sunitinib Monotherapy in Subjects With Previously Untreated, Advanced or Metastatic Renal Cell Carcinoma
Brief Title: Nivolumab Combined With Ipilimumab Versus Sunitinib in Previously Untreated Advanced or Metastatic Renal Cell Carcinoma (CheckMate 214)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-214; 2014-001750-42 (EudraCT Number)
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Advanced Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg (Experimental): Nivolumab 3 mg/kg combined with Ipilimumab 1 mg/kg solutions intravenously every 3 weeks for 4 doses then Nivolumab 3 mg/kg solutions intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm B: Sunitinib 50 mg (Active Comparator): Sunitinib 50 mg capsules by mouth once daily for 4 weeks then 2 weeks off, continuously until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  After completion of final analysis eligible participants may switch from receiving Sunitinib to receiving Nivolumab 3 mg/kg IV combined with Ipilimumab 1 mg/kg IV every 3 weeks for 4 doses then Nivolumab 240mg flat dose IV every 2 weeks
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Drug: Sunitinib

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558; Opdivo
Biological: Ipilimumab
  Other Names: Yervoy
Drug: Sunitinib
  Other Names: Sutent
  Arms: Arm B: Sunitinib 50 mg

SUMMARY:
The purpose of this study is to compare the objective response rate, progression free survival and the overall survival of Nivolumab combined with Ipilimumab to Sunitinib monotherapy in patients with previously untreated Renal Cell Cancer.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histological confirmation of renal cell carcinoma (RCC) with a clear-cell component
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (AJCC Stage IV) RCC
* No prior systemic therapy for RCC with the following exception:

  1. One prior adjuvant or neoadjuvant therapy for completely resectable RCC if such therapy did not include an agent that targets vascular endothelial growth factor (VEGF) or VEGF receptors and if recurrence occurred at least 6 months after the last dose of adjuvant or neoadjuvant therapy

     * Karnofsky Performance Status (KPS) of at least 70%
     * Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
     * Tumor tissue [formalin-fixed paraffin-embedded (FFPE) archival or recent acquisition] must be received by the central vendor (block or unstained slides) in order to randomize a subject to study treatment. (Note: Fine Needle Aspiration [FNA] and bone metastases samples are not acceptable for submission)

Exclusion Criteria:

* Any history of or current central nervous system (CNS) metastases. Baseline imaging of the brain is required within 28 days prior to randomization
* Prior systemic treatment with VEGF or VEGF receptor targeted therapy (including, but not limited to, Sunitinib, Pazopanib, Axitinib, Tivozanib, and Bevacizumab)
* Prior treatment with an anti-programmed death (PD)-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (>10 mg daily Prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger. Subjects with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll
* Any condition requiring systemic treatment with corticosteroids (>10 mg daily Prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses >10 mg daily Prednisone equivalents are permitted in the absence of active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1390 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2025-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (189):
- United States (37):
  - Local Institution - 0006, Duarte, California
  - Local Institution - 0057, La Jolla, California
  - Local Institution - 0044, Los Angeles, California
  - Local Institution - 0035, Los Angeles, California
  - Local Institution - 0067, Stanford, California
  - Local Institution - 0138, New Haven, Connecticut
  - Local Institution - 0034, Washington D.C., District of Columbia
  - Local Institution - 0049, Tampa, Florida
  - Local Institution - 0068, Atlanta, Georgia
  - Local Institution - 0038, Indianapolis, Indiana
  - Local Institution - 0042, Iowa City, Iowa
  - Local Institution - 0163, Fairway, Kansas
  - Local Institution - 0048, Baltimore, Maryland
  - Local Institution - 0004, Baltimore, Maryland
  - Local Institution - 0135, Boston, Massachusetts
  - Local Institution - 0110, Boston, Massachusetts
  - Local Institution - 0161, Boston, Massachusetts
  - Local Institution - 0173, Boston, Massachusetts
  - Local Institution - 0046, Ann Arbor, Michigan
  - Local Institution - 0043, Detroit, Michigan
  - Local Institution - 0036, Buffalo, New York
  - Local Institution - 0001, New York, New York
  - Local Institution - 0008, Charlotte, North Carolina
  - Local Institution - 0045, Durham, North Carolina
  - Local Institution - 0007, Cleveland, Ohio
  - Local Institution - 0164, Columbus, Ohio
  - Local Institution - 0039, Portland, Oregon
  - Local Institution - 0054, Allentown, Pennsylvania
  - Local Institution - 0005, Philadelphia, Pennsylvania
  - Local Institution - 0031, Pittsburgh, Pennsylvania
  - Local Institution - 0055, Charleston, South Carolina
  - Local Institution - 0159, Chattanooga, Tennessee
  - Local Institution - 0066, Nashville, Tennessee
  - Local Institution - 0056, Dallas, Texas
  - Local Institution - 0032, Dallas, Texas
  - Local Institution - 0003, Houston, Texas
  - Local Institution - 0041, Seattle, Washington
- Argentina (7):
  - Local Institution - 0099, Berazategui, Buenos Aires
  - Local Institution - 0098, Capital Federal, Buenos Aires
  - Local Institution - 0139, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution - 0095, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0096, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0097, CABA
  - Local Institution - 0100, Córdoba
- Australia (9):
  - Local Institution - 0073, Kogarah, New South Wales
  - Local Institution - 0070, Westmead, New South Wales
  - Local Institution - 0076, Herston, Queensland
  - Local Institution - 0075, Southport, Queensland
  - Local Institution - 0140, Elizabeth Vale, South Australia
  - Local Institution - 0072, Box Hill, Victoria
  - Local Institution - 0071, Clayton, Victoria
  - Local Institution - 0104, Nedlands, Western Australia
  - Local Institution - 0074, Murdoch
- Austria (3):
  - Local Institution - 0108, Linz
  - Local Institution - 0109, Vienna
  - Local Institution - 0107, Wels
- Belgium (2):
  - Local Institution - 0020, Ghent
  - Local Institution - 0019, Leuven
- Brazil (7):
  - Local Institution - 0152, Belo Horizonte, Minas Gerais
  - Local Institution - 0150, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0151, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0153, São Paulo, São Paulo
  - Local Institution - 0157, Rio de Janeiro
  - Local Institution - 0155, São Paulo
  - Local Institution - 0156, São Paulo
- Canada (8):
  - Local Institution - 0149, Calgary, Alberta
  - Local Institution - 0133, Edmonton, Alberta
  - Local Institution - 0182, Kelowna, British Columbia
  - Local Institution - 0128, Vancouver, British Columbia
  - Local Institution - 0131, Moncton, New Brunswick
  - Local Institution - 0172, Toronto, Ontario
  - Local Institution - 0148, Toronto, Ontario
  - Local Institution - 0132, Montreal, Quebec
- Chile (4):
  - Local Institution - 0101, Santiago, Santiago Metropolitan
  - Local Institution - 0102, Santiago, Santiago Metropolitan
  - Local Institution - 0144, Santiago, Santiago Metropolitan
  - Local Institution - 0103, Viña del Mar
- Colombia (3):
  - Local Institution - 0080, Bogotá
  - Local Institution - 0162, Medellín
  - Local Institution - 0081, Medellín
- Czechia (4):
  - Local Institution - 0050, Liberec, Liberecký kraj
  - Local Institution - 0053, Brno
  - Local Institution - 0051, Hradec Králové
  - Local Institution - 0052, Olomouc
- Denmark (3):
  - Local Institution - 0136, Aarhus N, Central Jutland
  - Local Institution - 0158, Herlev
  - Local Institution - 0137, Odense
- Finland (2):
  - Local Institution - 0027, Helsinki, Uusimaa
  - Local Institution - 0028, Tampere
- France (9):
  - Local Institution - 0170, Besançon
  - Local Institution - 0062, Bordeaux
  - Local Institution - 0169, La Roche-sur-Yon
  - Local Institution - 0060, Marseille
  - Local Institution - 0063, Saint-Herblain
  - Local Institution - 0065, Strasbourg
  - Local Institution - 0059, Toulouse
  - Local Institution - 0058, Villejuif
  - Local Institution - 0061, Paris, Île-de-France Region
- Germany (12):
  - Local Institution - 0125, Aachen
  - Local Institution - 0126, Erlangen
  - Local Institution - 0141, Frankfurt
  - Local Institution - 0147, Hamburg
  - Local Institution - 0142, Hanover
  - Local Institution - 0123, Heidelberg
  - Local Institution - 0127, Homburg
  - Local Institution - 0129, Jena
  - Local Institution - 0143, Magdeburg
  - Local Institution - 0124, München
  - Local Institution - 0146, Münster
  - Local Institution - 0130, Ulm
- Hungary (4):
  - Local Institution - 0184, Gyula, Bekes County
  - Local Institution - 0083, Budapest
  - Local Institution - 0082, Debrecen
  - Local Institution - 0084, Pécs
- Ireland (4):
  - Local Institution - 0015, Wilton, CORK
  - Local Institution - 0017, Dublin, Dublin
  - Local Institution - 0018, Dublin, Dublin
  - Local Institution - 0016, Dublin
- Israel (5):
  - Local Institution - 0120, Haifa
  - Local Institution - 0117, Kfar Saba
  - Local Institution - 0121, Petah Tikva
  - Local Institution - 0118, Ramat Gan
  - Local Institution - 0119, Ẕerifin
- Italy (7):
  - Local Institution - 0022, Arezzo
  - Local Institution - 0024, Meldola (fc)
  - Local Institution - 0023, Milan
  - Local Institution - 0064, Napoli
  - Local Institution - 0079, Padua
  - Local Institution - 0025, Pavia
  - Local Institution - 0026, Roma
- Japan (26):
  - Local Institution - 0192, Akita, Akita
  - Local Institution - 0209, Hirosaki, Aomori
  - Local Institution - 0187, Chiba, Chiba
  - Local Institution - 0196, Fukuoka, Fukuoka
  - Local Institution - 0188, Sapporo, Hokai-do
  - Local Institution - 0183, Sapporo, Hokkaido
  - Local Institution - 0206, Kobe, Hyōgo
  - Local Institution - 0205, Tsukuba, Ibaraki
  - Local Institution - 0200, Morioka, Iwate
  - Local Institution - 0186, Yokohama, Kanagawa
  - Local Institution - 0189, Kumamoto, Kumamoto
  - Local Institution - 0191, Kyoto, Kyoto
  - Local Institution - 0199, Niigata, Niigata
  - Local Institution - 0204, Okayama, Okayama-ken
  - Local Institution - 0190, Osakasayamashi, Osaka
  - Local Institution - 0201, Suita-shi, Osaka
  - Local Institution - 0208, Hamamatsu, Shizuoka
  - Local Institution - 0194, Tokushima, Tokushima
  - Local Institution - 0202, Bunkyo-ku, Tokyo
  - Local Institution - 0197, Bunkyo-ku, Tokyo
  - Local Institution - 0195, Bunkyo-ku, Tokyo
  - Local Institution - 0207, Koto-ku, Tokyo
  - Local Institution - 0185, Shinjuku-Ku, Tokyo
  - Local Institution - 0193, Shinjuku-ku, Tokyo
  - Local Institution - 0198, Tokyo
  - Local Institution - 0203, Yamagata
- Mexico (4):
  - Local Institution - 0168, Mexico City, Mexico City
  - Local Institution - 0171, Monterrey, Nuevo León
  - Local Institution - 0175, Querétaro City, Querétaro
  - Local Institution - 0167, Oaxaca City
- Netherlands (3):
  - Local Institution - 0029, Amsterdam, North Holland
  - Local Institution - 0040, Groningen
  - Local Institution - 0030, Nijmegen
- Poland (3):
  - Local Institution - 0093, Krakow
  - Local Institution - 0112, Poznan
  - Local Institution - 0106, Wroclaw
- South Korea (3):
  - Local Institution - 0178, Seoul
  - Local Institution - 0177, Seoul
  - Local Institution - 0176, Seoul
- Spain (7):
  - Local Institution - 0089, Barcelona
  - Local Institution - 0088, Barcelona
  - Local Institution - 0086, Madrid
  - Local Institution - 0085, Madrid
  - Local Institution - 0087, Madrid
  - Local Institution - 0111, Oviedo
  - Local Institution - 0090, Seville
- Local Institution - 0134, Stockholm, Sweden
- Taiwan (3):
  - Local Institution - 0179, Taipei
  - Local Institution - 0180, Taipei
  - Local Institution - 0181, Taoyuan District
- Turkey (Türkiye) (3):
  - Local Institution - 0115, Ankara
  - Local Institution - 0114, Antalya
  - Local Institution - 0122, Istanbul
- United Kingdom (6):
  - Local Institution - 0010, London, Greater London
  - Local Institution - 0009, Glasgow, Lanarkshire
  - Local Institution - 0077, London
  - Local Institution - 0021, Manchester
  - Local Institution - 0011, Northwood
  - Local Institution - 0012, Swansea

REFERENCES:
- [Derived] Mantia CM, Jegede OA, Plimack ER, Powles T, Motzer RJ, Tannir NM, Lee CH, Tomita Y, Voss MH, Choueiri TK, Rini BI, Hammers HJ, Escudier B, Albiges L, Rosenblatt L, Atkins MB, Regan MM, McDermott DF. Treatment-free survival and partitioned survival analysis of patients with advanced renal cell carcinoma treated with nivolumab plus ipilimumab versus sunitinib: 5-year update of CheckMate 214. J Immunother Cancer. 2024 Jul 25;12(7):e009495. doi: 10.1136/jitc-2024-009495. PMID 39060019
- [Derived] Cella D, Choueiri TK, Hamilton M, Blum SI, Ivanescu C, Karu K, Ejzykowicz F, Motzer RJ. The Relationship Between Health-Related Quality of Life and Overall Survival in Patients With Advanced Renal Cell Carcinoma in CheckMate 214. Oncologist. 2024 Jun 3;29(6):511-518. doi: 10.1093/oncolo/oyae003. PMID 38280218
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Rini BI, Signoretti S, Choueiri TK, McDermott DF, Motzer RJ, George S, Powles T, Donskov F, Tykodi SS, Pal SK, Gupta S, Lee CW, Jiang R, Tannir NM. Long-term outcomes with nivolumab plus ipilimumab versus sunitinib in first-line treatment of patients with advanced sarcomatoid renal cell carcinoma. J Immunother Cancer. 2022 Dec;10(12):e005445. doi: 10.1136/jitc-2022-005445. PMID 36549781
- [Derived] Motzer RJ, McDermott DF, Escudier B, Burotto M, Choueiri TK, Hammers HJ, Barthelemy P, Plimack ER, Porta C, George S, Powles T, Donskov F, Gurney H, Kollmannsberger CK, Grimm MO, Barrios C, Tomita Y, Castellano D, Grunwald V, Rini BI, McHenry MB, Lee CW, McCarthy J, Ejzykowicz F, Tannir NM. Conditional survival and long-term efficacy with nivolumab plus ipilimumab versus sunitinib in patients with advanced renal cell carcinoma. Cancer. 2022 Jun 1;128(11):2085-2097. doi: 10.1002/cncr.34180. Epub 2022 Apr 5. PMID 35383908
- [Derived] Labriola MK, George DJ. Setting a new standard for long-term survival in metastatic kidney cancer. Cancer. 2022 Jun 1;128(11):2058-2060. doi: 10.1002/cncr.34177. Epub 2022 Apr 5. No abstract available. PMID 35383907
- [Derived] Albiges L, Tannir NM, Burotto M, McDermott D, Plimack ER, Barthelemy P, Porta C, Powles T, Donskov F, George S, Kollmannsberger CK, Gurney H, Grimm MO, Tomita Y, Castellano D, Rini BI, Choueiri TK, Leung D, Saggi SS, Lee CW, McHenry MB, Motzer RJ. First-line Nivolumab plus Ipilimumab Versus Sunitinib in Patients Without Nephrectomy and With an Evaluable Primary Renal Tumor in the CheckMate 214 Trial. Eur Urol. 2022 Mar;81(3):266-271. doi: 10.1016/j.eururo.2021.10.001. Epub 2021 Nov 5. PMID 34750035
- [Derived] Albiges L, Tannir NM, Burotto M, McDermott D, Plimack ER, Barthelemy P, Porta C, Powles T, Donskov F, George S, Kollmannsberger CK, Gurney H, Grimm MO, Tomita Y, Castellano D, Rini BI, Choueiri TK, Saggi SS, McHenry MB, Motzer RJ. Nivolumab plus ipilimumab versus sunitinib for first-line treatment of advanced renal cell carcinoma: extended 4-year follow-up of the phase III CheckMate 214 trial. ESMO Open. 2020 Nov;5(6):e001079. doi: 10.1136/esmoopen-2020-001079. PMID 33246931
- [Derived] Motzer RJ, Escudier B, McDermott DF, Aren Frontera O, Melichar B, Powles T, Donskov F, Plimack ER, Barthelemy P, Hammers HJ, George S, Grunwald V, Porta C, Neiman V, Ravaud A, Choueiri TK, Rini BI, Salman P, Kollmannsberger CK, Tykodi SS, Grimm MO, Gurney H, Leibowitz-Amit R, Geertsen PF, Amin A, Tomita Y, McHenry MB, Saggi SS, Tannir NM. Survival outcomes and independent response assessment with nivolumab plus ipilimumab versus sunitinib in patients with advanced renal cell carcinoma: 42-month follow-up of a randomized phase 3 clinical trial. J Immunother Cancer. 2020 Jul;8(2):e000891. doi: 10.1136/jitc-2020-000891. PMID 32661118
- [Derived] Ambavane A, Yang S, Atkins MB, Rao S, Shah A, Regan MM, McDermott DF, Michaelson MD. Clinical and economic outcomes of treatment sequences for intermediate- to poor-risk advanced renal cell carcinoma. Immunotherapy. 2020 Jan;12(1):37-51. doi: 10.2217/imt-2019-0199. Epub 2020 Jan 29. PMID 31992108
- [Derived] Tomita Y, Kondo T, Kimura G, Inoue T, Wakumoto Y, Yao M, Sugiyama T, Oya M, Fujii Y, Obara W, Motzer RJ, Uemura H. Nivolumab plus ipilimumab versus sunitinib in previously untreated advanced renal-cell carcinoma: analysis of Japanese patients in CheckMate 214 with extended follow-up. Jpn J Clin Oncol. 2020 Jan 24;50(1):12-19. doi: 10.1093/jjco/hyz132. PMID 31633185
- [Derived] Motzer RJ, Rini BI, McDermott DF, Aren Frontera O, Hammers HJ, Carducci MA, Salman P, Escudier B, Beuselinck B, Amin A, Porta C, George S, Neiman V, Bracarda S, Tykodi SS, Barthelemy P, Leibowitz-Amit R, Plimack ER, Oosting SF, Redman B, Melichar B, Powles T, Nathan P, Oudard S, Pook D, Choueiri TK, Donskov F, Grimm MO, Gurney H, Heng DYC, Kollmannsberger CK, Harrison MR, Tomita Y, Duran I, Grunwald V, McHenry MB, Mekan S, Tannir NM; CheckMate 214 investigators. Nivolumab plus ipilimumab versus sunitinib in first-line treatment for advanced renal cell carcinoma: extended follow-up of efficacy and safety results from a randomised, controlled, phase 3 trial. Lancet Oncol. 2019 Oct;20(10):1370-1385. doi: 10.1016/S1470-2045(19)30413-9. Epub 2019 Aug 16. PMID 31427204
- [Derived] Cella D, Grunwald V, Escudier B, Hammers HJ, George S, Nathan P, Grimm MO, Rini BI, Doan J, Ivanescu C, Paty J, Mekan S, Motzer RJ. Patient-reported outcomes of patients with advanced renal cell carcinoma treated with nivolumab plus ipilimumab versus sunitinib (CheckMate 214): a randomised, phase 3 trial. Lancet Oncol. 2019 Feb;20(2):297-310. doi: 10.1016/S1470-2045(18)30778-2. Epub 2019 Jan 15. PMID 30658932
- [Derived] Motzer RJ, Tannir NM, McDermott DF, Aren Frontera O, Melichar B, Choueiri TK, Plimack ER, Barthelemy P, Porta C, George S, Powles T, Donskov F, Neiman V, Kollmannsberger CK, Salman P, Gurney H, Hawkins R, Ravaud A, Grimm MO, Bracarda S, Barrios CH, Tomita Y, Castellano D, Rini BI, Chen AC, Mekan S, McHenry MB, Wind-Rotolo M, Doan J, Sharma P, Hammers HJ, Escudier B; CheckMate 214 Investigators. Nivolumab plus Ipilimumab versus Sunitinib in Advanced Renal-Cell Carcinoma. N Engl J Med. 2018 Apr 5;378(14):1277-1290. doi: 10.1056/NEJMoa1712126. Epub 2018 Mar 21. PMID 29562145
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 1390 patients were enrolled in the study. Of these, 1096 were randomized. Of those randomized, 1082 received treatment (547 with Nivo+Ipi and 535 with Sunitinib). 240 patients who were not randomized because they no longer met study criteria, 24 withdrew consent, 4 for Adverse Events, 4 for Death, 4 for Poor Compliance, and 18 other.
Groups:
- Nivolumab + Ipilimumab: Nivolumab 3 mg/kg combined with Ipilimumab 1 mg/kg solutions intravenously every 3 weeks for 4 doses then Nivolumab 3 mg/kg solutions intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
- Sunitinib: Sunitinib 50 mg capsules by mouth once daily for 4 weeks then 2 weeks off, continuously until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends After completion of final analysis eligible participants may switch from receiving Sunitinib to receiving Nivolumab 3 mg/kg IV combined with Ipilimumab 1 mg/kg IV every 3 weeks for 4 doses then Nivolumab 240mg flat dose IV every 2 weeks
Period: Overall Study
Arm/Group | Nivolumab + Ipilimumab | Sunitinib
Started (Started = Randomized) | 550 | 546
Received Treatment | 547 | 535
Completed (Completed = Continuing in the Treatment Period) | 128 | 97
Not Completed | 422 | 449
Not completed — Disease progression | 229 | 297
Not completed — Study Drug Toxicity | 134 | 63
Not completed — Death | 1 | 1
Not completed — AE unrelated to Study drug | 32 | 31
Not completed — Participant's request to discontinue | 10 | 21
Not completed — Participant withdrew Consent | 8 | 15
Not completed — Lost to Follow-up | 1 | 2
Not completed — Maximum Clinical Benefit | 5 | 8
Not completed — Poor/Non-Compliance | 0 | 3
Not completed — Pregnancy | 1 | 0
Not completed — other | 0 | 8
Not completed — No longer meets Study Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + Ipilimumab | Sunitinib | Total
Number analyzed (Participants) | 550 | 546 | 1096
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All Randomized
  Years | 61.1 (9.76) | 60.7 (10.10) | 60.9 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All Randomized Participants
  Participants
    Female | 137 | 151 | 288
    Male | 413 | 395 | 808
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 17 | 29
  Not Hispanic or Latino | 264 | 253 | 517
  Unknown or Not Reported | 274 | 276 | 550
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: All Randomized Participants
  Participants
    White | 486 | 483 | 969
    Black or African American | 7 | 6 | 13
    Asian | 46 | 47 | 93
    American Indian or Alaska Native | 0 | 0 | 0
    Native Hawaiian or Pacific Islander | 0 | 0 | 0
    Other | 10 | 10 | 20
    Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Objective Response Rate(ORR) in Intermediate/Poor Risk Participants Per IRRC Using RECIST v1.1
Description: ORR was defined as the proportion of randomized subjects who achieved a best response of complete response (CR) or partial response (PR) using the RECIST v1.1 criteria based on IRRC assessment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), greater than or equal to 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From first dose until date of documented disease progression or subsequent therapy, whichever occurs first (assessed up to June 2017, approximately 31 months)
Population: All Intermediate/Poor-Risk Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab + Ipilimumab | Sunitinib
Number analyzed (Participants) | 425 | 422
percentage of participants | 41.6 [36.9 to 46.5] | 26.5 [22.4 to 31.0]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Sunitinib; Test type: Superiority; p < 0.0001, DerSimonian and Laird Test; Stratified Difference = 16.0, 95% CI 2-sided [9.8 to 22.2]

2. Primary Outcome: Overall Survival (OS) in Intermediate/Poor-Risk Participants With Previously Untreated Metastatic Renal Cell Carcinoma (mRCC)
Description: OS was defined as the time from randomization to the date of death from any cause. Survival time was censored at the date of last contact ("last known alive date") for subjects who were alive.
Time Frame: From the date of randomization to the date of death (assessed up to June 2017, approximately 31 months)
Population: All Intermediate/Poor-Risk Participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Ipilimumab | Sunitinib
Number analyzed (Participants) | 425 | 422
months | NA [28.16 to NA] — The median for Overall Survival and Upper Limit have not been reached. There were an insufficient number of participants with events. | 25.95 [22.08 to NA] — The median for Overall Survival and Upper Limit have not been reached. There were an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Sunitinib; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.63, 99.8% CI 2-sided [0.44 to 0.89]

3. Primary Outcome: Progression-Free Survival (PFS) in Intermediate/Poor-Risk Participants With Previously Untreated Metastatic Renal Cell Carcinoma (mRCC)
Description: PFS was defined as the time between the date of randomization and the first date of documented progression, as determined by the IRRC (as per RECIST 1.1 criteria), or death due to any cause, whichever occurred first. Subsequent therapy included anticancer therapy, tumor directed radiotherapy, or tumor directed surgery. Subjects who died without a reported progression were considered to have progressed on the date of their death.
Time Frame: From date of first dose to date of documented disease progression or death due to any cause, whichever occurs first (assessed up to June 2017, approximately 31 months)
Population: All Intermediate/Poor-Risk Participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Ipilimumab | Sunitinib
Number analyzed (Participants) | 425 | 422
months | 11.56 [8.71 to 15.51] | 8.38 [7.03 to 10.81]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Sunitinib; Test type: Superiority; p = 0.0331, Log Rank; Hazard Ratio (HR) = 0.82, 99.1% CI 2-sided [0.64 to 1.05]

4. Secondary Outcome: Investigator-assessed Objective Response Rate(ORR) in Any Risk Participants Per IRRC Using RECIST v1.1
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All Randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab + Ipilimumab | Sunitinib
Number analyzed (Participants) | 550 | 546
percentage of participants | 38.7 [34.6 to 42.9] | 32.2 [28.3 to 36.3]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Sunitinib; Test type: Superiority; p = 0.0191, DerSimonian and Laird Test; Stratified Difference = 7.2, 95% CI 2-sided [1.8 to 12.7]

5. Secondary Outcome: Overall Survival (OS) in Any Risk Participants With Previously Untreated Metastatic Renal Cell Carcinoma (mRCC)
Description: Overall survival is defined as the time from randomization to the date of death from any cause. For subjects that are alive, their survival time will be censored at the date of last contact ("last known alive date"). Overall survival will be censored for subjects at the date of randomization if they were randomized but had no follow-up. Survival follow-up will be conducted every 3 months after subject's off-treatment date.
Time Frame: From the date of randomization to the date of death (assessed up to June 2017, approximately 31 months)
Population: All Randomized
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Ipilimumab | Sunitinib
Number analyzed (Participants) | 550 | 546
months | NA [NA to NA] — The median for Overall Survival, Lower limit, and Upper Limit have not been reached. There were an insufficient number of participants with events. | 32.92 [NA to NA] — The Lower Limit and Upper Limit have not been reached. With only 1 participant at that time point, the variance is not estimable and so the Confidence Intervals were N/A.
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Sunitinib; Test type: Superiority; p = 0.0003, Log Rank; Hazard Ratio (HR) = 0.68, 99.8% CI 2-sided [0.49 to 0.95]

6. Secondary Outcome: Progression-Free Survival (PFS) in Any Risk Participants With Previously Untreated Metastatic Renal Cell Carcinoma (mRCC)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: All Randomized
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Ipilimumab | Sunitinib
Number analyzed (Participants) | 550 | 546
months | 12.42 [9.89 to 16.53] | 12.32 [9.79 to 15.24]
Statistical Analysis 1: Comparison: Nivolumab + Ipilimumab vs Sunitinib; Test type: Superiority; p = 0.8498, Log Rank; Hazard Ratio (HR) = 0.98, 99.1% CI 2-sided [0.79 to 1.23]

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after last dose of study therapy (assessed up to June 2017, approximately 31 months)
Arm/Group | Nivolumab + Ipilimumab | Sunitinib
All-Cause Mortality (participants affected / at risk) | 159/547 | 202/535
Serious Adverse Events (participants affected / at risk) | 305/547 | 213/535
Other Adverse Events (participants affected / at risk) | 530/547 | 522/535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=547) | Sunitinib (N=535)
Anaemia (Blood and lymphatic system disorders) | 6 | 7
Autoimmune neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Splenic lesion (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 3 | 2
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 3
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 6 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 10 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 2 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Autoimmune hypothyroidism (Endocrine disorders) | 1 | 0
Basedow's disease (Endocrine disorders) | 2 | 0
Goitre (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 3 | 0
Hypophysitis (Endocrine disorders) | 14 | 0
Hypopituitarism (Endocrine disorders) | 2 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 2 | 0
Steroid withdrawal syndrome (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 3 | 0
Diplopia (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 1 | 0
Inflammation of lacrimal passage (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 10 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 3
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 4
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 4
Asthenia (General disorders) | 1 | 4
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 2
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 5
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 4 | 4
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 2
Mucosal inflammation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 18 | 9
Sudden death (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 3 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Autoimmune disorder (Immune system disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 3 | 0
Contrast media reaction (Immune system disorders) | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 3 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Herpes zoster disseminated (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 2
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Lung abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 2 | 1
Meningitis aseptic (Infections and infestations) | 2 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 17 | 8
Pulmonary sepsis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 6
Septic shock (Infections and infestations) | 2 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 6 | 0
Urosepsis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Drug administration error (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 9 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 5 | 1
Blood potassium increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Pancreatic enzymes increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 4
Transaminases increased (Investigations) | 3 | 0
Troponin increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 31
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 3 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cervical cord compression (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 1
Iiird nerve paralysis (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 2 | 1
Thecal sac compression (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Visual field defect (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Device breakage (Product Issues) | 1 | 0
Confusional state (Psychiatric disorders) | 6 | 0
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 8 | 8
Autoimmune nephritis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 8
Micturition urgency (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 3
Renal impairment (Renal and urinary disorders) | 1 | 2
Renal injury (Renal and urinary disorders) | 2 | 0
Renal mass (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 15 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Immobile (Social circumstances) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 3
Embolism (Vascular disorders) | 2 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 4 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Subclavian vein occlusion (Vascular disorders) | 1 | 0
Vein rupture (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=547) | Sunitinib (N=535)
Anaemia (Blood and lymphatic system disorders) | 71 | 108
Leukopenia (Blood and lymphatic system disorders) | 1 | 31
Neutropenia (Blood and lymphatic system disorders) | 3 | 73
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 98
Hyperthyroidism (Endocrine disorders) | 63 | 16
Hypothyroidism (Endocrine disorders) | 94 | 144
Vision blurred (Eye disorders) | 28 | 10
Abdominal distension (Gastrointestinal disorders) | 14 | 27
Abdominal pain (Gastrointestinal disorders) | 69 | 76
Abdominal pain upper (Gastrointestinal disorders) | 26 | 44
Constipation (Gastrointestinal disorders) | 93 | 94
Diarrhoea (Gastrointestinal disorders) | 198 | 310
Dry mouth (Gastrointestinal disorders) | 35 | 37
Dyspepsia (Gastrointestinal disorders) | 29 | 112
Flatulence (Gastrointestinal disorders) | 7 | 31
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 67
Haemorrhoids (Gastrointestinal disorders) | 12 | 27
Nausea (Gastrointestinal disorders) | 161 | 230
Oral pain (Gastrointestinal disorders) | 2 | 30
Stomatitis (Gastrointestinal disorders) | 29 | 152
Toothache (Gastrointestinal disorders) | 9 | 27
Vomiting (Gastrointestinal disorders) | 108 | 148
Asthenia (General disorders) | 88 | 99
Chest pain (General disorders) | 23 | 27
Chills (General disorders) | 31 | 42
Fatigue (General disorders) | 246 | 291
Influenza like illness (General disorders) | 46 | 27
Malaise (General disorders) | 12 | 28
Mucosal inflammation (General disorders) | 18 | 156
Oedema peripheral (General disorders) | 75 | 66
Pain (General disorders) | 33 | 45
Pyrexia (General disorders) | 126 | 85
Upper respiratory tract infection (Infections and infestations) | 34 | 35
Urinary tract infection (Infections and infestations) | 29 | 24
Viral upper respiratory tract infection (Infections and infestations) | 46 | 21
Alanine aminotransferase increased (Investigations) | 63 | 60
Amylase increased (Investigations) | 76 | 42
Aspartate aminotransferase increased (Investigations) | 69 | 57
Blood alkaline phosphatase increased (Investigations) | 32 | 24
Blood creatinine increased (Investigations) | 65 | 49
Blood thyroid stimulating hormone increased (Investigations) | 12 | 32
Lipase increased (Investigations) | 96 | 65
Neutrophil count decreased (Investigations) | 5 | 40
Platelet count decreased (Investigations) | 9 | 76
Weight decreased (Investigations) | 47 | 41
White blood cell count decreased (Investigations) | 6 | 41
Decreased appetite (Metabolism and nutrition disorders) | 114 | 156
Dehydration (Metabolism and nutrition disorders) | 28 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 54 | 23
Hyperkalaemia (Metabolism and nutrition disorders) | 36 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 | 32
Hyponatraemia (Metabolism and nutrition disorders) | 33 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 122 | 83
Back pain (Musculoskeletal and connective tissue disorders) | 87 | 89
Muscle spasms (Musculoskeletal and connective tissue disorders) | 34 | 28
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 36 | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 64 | 34
Pain in extremity (Musculoskeletal and connective tissue disorders) | 62 | 76
Dizziness (Nervous system disorders) | 61 | 61
Dysgeusia (Nervous system disorders) | 40 | 185
Headache (Nervous system disorders) | 102 | 120
Paraesthesia (Nervous system disorders) | 33 | 29
Anxiety (Psychiatric disorders) | 29 | 21
Insomnia (Psychiatric disorders) | 58 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 144 | 125
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 | 28
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 95 | 92
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 75
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 26 | 40
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 27
Dry skin (Skin and subcutaneous tissue disorders) | 55 | 53
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 32
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 | 237
Pruritus (Skin and subcutaneous tissue disorders) | 180 | 58
Rash (Skin and subcutaneous tissue disorders) | 139 | 84
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 55 | 28
Skin discolouration (Skin and subcutaneous tissue disorders) | 3 | 27
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 45
Hypertension (Vascular disorders) | 52 | 230

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT02231749/Prot_001.pdf
  • Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02231749/SAP_000.pdf